CLINICAL TRIAL: NCT00530816
Title: An Open-label, Single-arm, Phase 2 Study of Carfilzomib in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Phase 2 Study of Carfilzomib in Relapsed Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PX-171-004
Record Dates: First submitted 2007-09-14; First posted 2007-09-18 (Estimated); Results first posted 2015-12-03 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-04

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — carfilzomib; WW Domain-Containing Oxidoreductase

ARMS (1):
- Carfilzomib (Experimental): Participants received carfilzomib 20 mg/m² intravenous (IV) injection on Days 1, 2, 8, 9, 15, and 16, in 28-day treatment cycles for a maximum of 12 cycles.
  Starting with Amendment 3, if all doses in Cycle 1 were well-tolerated the dose was escalated to 27 mg/m² IV for subsequent cycles.
  Interventions: Drug: carfilzomib

INTERVENTIONS:
Drug: carfilzomib — Intravenous (IV) injection over 2 to 10 minutes twice weekly for three weeks followed by 12 days of rest.
  Other Names: PR-171; PR171; Kyprolis® (carfilzomib) for Injection

SUMMARY:
To evaluate the best overall response rate, safety and tolerability of carfilzomib in patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
Two groups of patients with multiple myeloma were initially studied: bortezomib-naïve and bortezomib-treated. Following Amendment 2, only bortezomib-naïve patients were enrolled. Study results were reported in 2 parts, depending on whether a patient received prior bortezomib.

ELIGIBILITY:
Inclusion Criteria:

Disease Related

* Multiple myeloma
* Subjects must have measurable disease, defined as one or more of the following:

  * Serum M-protein ≥ 1 g/dL
  * Urine M-protein ≥ 200 mg/24 hours
* Subjects must have been responsive (i.e., achieve a minimal response [MR] or better) to standard, first line therapy
* Relapsed and/or refractory or progressive disease after at least one, but no more than three, prior therapeutic treatments or regimens for multiple myeloma. Refractory disease is defined as ≤ 25% response or progression during therapy or within 60 days after completion of therapy. Induction therapy and stem cell transplant will be considered as one regimen

Demographic

* Males and females ≥18 years of age
* Life expectancy of more than three months
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2

Laboratory

* Adequate hepatic function, with bilirubin < 2.0 times the upper limit of normal, and aspartate aminotransferase (AST) and alanine aminotransferase (ALT) of < 3.0 times the upper limit of normal
* Uric acid, if elevated, must be corrected to within laboratory normal range prior to dosing
* Total white blood cell (WBC) count ≥ 2,000/mm³, absolute neutrophil count > 1,000/mm³, hemoglobin ≥ 8.0 g/dL, and platelet count > 50,000/mm³
* Subjects should be platelet transfusion independent
* Screening absolute neutrophil count (ANC) should be independent of granulocyte colony stimulating factor (G-CSF) or granulocyte macrophage colony stimulating factor (GM-CSF) support for ≥ 1 week and of pegylated G-CSF for ≥ 2 weeks
* Subjects may receive red blood cell (RBC) transfusion or receive supportive care such as erythropoietin and darbepoetin in accordance with institutional guidelines
* Calculated or measured creatinine clearance of ≥ 30 mL/minute, calculated using the formula of Cockcroft and Gault [(140 - Age) X Mass (kg) / (72 X Creatinine mg/dL)]. Multiply result by 0.85 if female.
* Serum creatinine ≤ 2 mg/dL

Ethical / Other

* Written informed consent in accordance with federal, local, and institutional guidelines
* Female subjects of child-bearing potential must have a negative serum pregnancy test within seven days of the first dose and agree to use dual methods of contraception during and for 3 months following last dose of drug. Post menopausal females (> 45 years old and without menses for > 1 year) and surgically sterilized females are exempt from a pregnancy test. Male subjects must use an effective barrier method of contraception during study and for 3 months following the last dose if sexually active with a female of child-bearing potential.
* Subjects must be able to receive outpatient treatment and laboratory monitoring at the institute that administers agent.

Exclusion Criteria:

Disease Related

* Multiple Myeloma Immunoglobulin M (IgM)
* Subjects previously treated with any proteasome inhibitor (for Part 2 Proteasome Inhibitor - Naïve only, criteria added at Amendment 2)
* Subjects must not be primary refractory to standard first-line therapy
* Subjects with non-secretory multiple myeloma, defined as < 1 g/dL M-protein in serum, < 200 mg/24 hour M-protein in urine
* Subjects with disease measurable only by serum free light chain (SFLC) analysis
* Glucocorticoid therapy (prednisone >10 mg/day orally or equivalent) within the last three weeks
* POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes)
* Plasma cell leukemia
* Chemotherapy with approved or investigative anticancer therapeutics, including steroid therapy, within the three weeks prior to first dose
* Radiation therapy or immunotherapy in the previous four weeks; localized radiation therapy within 1 week prior to first dose
* Participation in an investigational therapeutic study within three weeks or within five drug half-lives (t1/2) prior to first dose, whichever time is greater
* Prior treatment with carfilzomib

Concurrent Conditions

* Major surgery within three weeks before Day 1
* Congestive heart failure (New York Heart Association class III to IV), symptomatic ischemia, conduction abnormalities uncontrolled by conventional intervention, or myocardial infarction in the previous six months
* Acute active infection requiring systemic antibiotics, antivirals or antifungals within 2 weeks prior to first dose
* Known or suspected human immunodeficiency (HIV) infection or subjects who are HIV seropositive
* Active hepatitis A, B, or C infection
* Non-hematologic malignancy within the past three years except a) adequately treated basal cell or squamous cell skin cancer, b) carcinoma in situ of the cervix, or c) prostate cancer < Gleason Grade 6 with stable prostate-specific antigen (PSA)
* Subjects with treatment related myelodysplastic syndrome
* Significant neuropathy (Grade 3, 4 or Grade 2 with pain) at the time of study initiation
* Subjects with known contraindication to receiving allopurinol
* Subjects in whom the required program of oral and intravenous fluid hydration is contraindicated, e.g., due to pre-existing pulmonary, cardiac, or renal impairment
* Subjects with known or suspected amyloidosis Subjects with pleural effusions requiring thoracentesis or ascites requiring paracentesis
* Any clinically significant medical disease or condition that, in the Investigator's opinion, may interfere with protocol adherence or a subject's ability to give informed consent

Ethical / Other

* Female subjects who are pregnant or lactating
* Serious psychiatric or medical conditions that could interfere with treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2007-09; Primary Completion 2013-01 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (30):
- United States (26):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Tower Cancer Research Foundation, Beverly Hills, California
  - Therapeutic Research Institute of Orange County, Laguna Hills, California
  - Rocky Mountain Blood and Marrow Transplant Program, Denver, Colorado
  - Oncology & Hematology Assoc. of W. Broward, Tamarac, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Orchard Research, Skokie, Illinois
  - University of Kentucky College of Medicine, Lexington, Kentucky
  - Montgomery Cancer Center, Mount Sterling, Kentucky
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Jackson Oncology Associates, Jackson, Mississippi
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - St. Vincent's Comprehensive Cancer Center, New York, New York
  - Summa Health System, Akron, Ohio
  - Gabrail Cancer Center, Canton, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Dayton Clinical Oncology Program, Dayton, Ohio
  - Signal Point Clinical Research Center, LLC, Middletown, Ohio
  - Harrington Cancer Center, Amarillo, Texas
  - Texas Oncology Cancer Center, Austin, Texas
  - MD Anderson Cancer Center, Houston, Texas
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - University of Alberta Cross Cancer Institute, Edmonton, Alberta
  - University of Toronto Princess Margaret Hospital, Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec

REFERENCES:
- [Derived] Vij R, Wang M, Kaufman JL, Lonial S, Jakubowiak AJ, Stewart AK, Kukreti V, Jagannath S, McDonagh KT, Alsina M, Bahlis NJ, Reu FJ, Gabrail NY, Belch A, Matous JV, Lee P, Rosen P, Sebag M, Vesole DH, Kunkel LA, Wear SM, Wong AF, Orlowski RZ, Siegel DS. An open-label, single-arm, phase 2 (PX-171-004) study of single-agent carfilzomib in bortezomib-naive patients with relapsed and/or refractory multiple myeloma. Blood. 2012 Jun 14;119(24):5661-70. doi: 10.1182/blood-2012-03-414359. Epub 2012 May 3. PMID 22555973

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled patients with multiple myeloma (MM) who had relapsed or refractory disease after at least 1 but no more than 3 prior therapeutic treatments or regimens. The first patient enrolled on 24 September 2007; the last patient was enrolled and received carfilzomib on 28 May 2009.
Pre-assignment Details: Two groups of patients with MM were initially studied: bortezomib-treated (Part 1) and bortezomib-naïve (Part 2). Following Amendment 2, only bortezomib-naïve patients were enrolled. With Amendment 3, a new cohort of "stepped up" dosing was added to the trial. Study results were analyzed in 2 parts, based on previous bortezomib treatment.
Groups:
- Part 1: Carfilzomib 20 mg/m²: Participants previously treated with bortezomib received carfilzomib 20 mg/m² intravenous (IV) injection on Days 1, 2, 8, 9, 15, and 16, in 28-day treatment cycles for a maximum of 12 cycles.
- Part 2: Carfilzomib 20 mg/m²: Participants not previously treated with bortezomib received carfilzomib 20 mg/m² IV injection on Days 1, 2, 8, 9, 15, and 16, in 28-day treatment cycles for a maximum of 12 cycles.
- Part 2: Carfilzomib 20/27 mg/m²: Participants not previously treated with bortezomib received carfilzomib 20 mg/m² IV on Days 1, 2, 8, 9, 15, and 16 of Cycle 1. If all doses were well-tolerated the dose was escalated to 27 mg/m² IV on Days 1, 2, 8, 9, 15, and 16 of subsequent cycles, for up to 12 cycles.
Period: Overall Study
Arm/Group | Part 1: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20/27 mg/m²
Started | 35 | 59 | 70
Completed | 9 | 17 | 29
Not Completed | 26 | 42 | 41
Not completed — Progressive Disease | 16 | 24 | 24
Not completed — Adverse Event | 6 | 13 | 7
Not completed — Other | 3 | 3 | 4
Not completed — Withdrawal by Subject | 1 | 2 | 6

BASELINE CHARACTERISTICS:
Population: Safety Population: All patients enrolled on study and who received at least 1 dose of carfilzomib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20/27 mg/m² | Total
Number analyzed (Participants) | 35 | 59 | 70 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 21 | 29 | 31 | 81
  >=65 years | 14 | 30 | 39 | 83
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 27 | 26 | 70
  Male | 18 | 32 | 44 | 94
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status is used by doctors and researchers to assess how a participants disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active; 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, no self-care, confined to bed or chair; 5 = Death.
  participants
    0 (Fully Active) | 15 | 29 | 23 | 67
    1 (Restrictive but ambulatory) | 18 | 27 | 42 | 87
    2 (Ambulatory but unable to work) | 1 | 3 | 5 | 9
    Missing | 1 | 0 | 0 | 1
Measurable Disease Category [Number; unit: participants] — Measurable disease categories defined as:
  SPEP: Serum M-protein ≥ 1 g/dL by serum protein electrophoresis (SPEP);
  UPEP: Urine M-protein ≥ 200 mg/24 hour by urine protein electrophoresis (UPEP);
  SPEP and UPEP: M-protein levels ≥ 1 g/dL in serum and ≥ 200 mg/24 hours;
  SFLC Only: Detectable using serum free light chain (SFLC) assay only (participants enrolled prior to Amendment 2);
  IgA only: For patients with immunoglobulin A (IgA) myeloma for whom SPEP is considered unreliable, quantitative immunoglobulin (e.g. nephelometry or turbidometry) was performed.
  participants
    SPEP and UPEP | 3 | 6 | 11 | 20
    SPEP | 22 | 39 | 47 | 108
    UPEP | 6 | 6 | 10 | 22
    SFLC Only | 4 | 6 | 1 | 11
    IgA, by Immunoglobulin Assay Only | 0 | 2 | 0 | 2
    Missing | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rate (ORR) in the Response Evaluable Subset Population
Description: ORR is defined as the percentage of patients who achieved a best response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR) determined by Independent Review Committee (IRC). Responses were assessed according to International Uniform Response Criteria for Multiple Myeloma, documented by 2 consecutive assessments made at any time before the start of new therapy.
  sCR: CR as defined below plus normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunofluorescence.
  CR: absence of M-protein in serum and urine by immunofixation, disappearance of any soft tissue plasmacytomas, and ≤5% plasma cells in bone marrow.
  VGPR: serum and urine M-proteins detectable by immunofixation but not by electrophoresis or a ≥ 90% reduction in serum M-protein with urine M-protein level < 100 mg/24 hours.
  PR: ≥ 50% reduction of serum M-protein and in urine of ≥ 90% or to < 200 mg per 24 hours.
Time Frame: Disease response was assessed on Day 15 of Cycle 1, Day 1 of Cycles 2 through 12, and at End of Study, 30 days after last dose. Median duration of treatment was 100 days for Part 1 and 170 days for Part 2 participants.
Population: The Response Evaluable Subset population consists of all treated patients with measurable disease at Baseline as assessed by M-protein or by quantitative serum Ig for certain patients with IgA myeloma, and with a baseline and at least 1 post-baseline disease assessment.
  Patients whose disease was only measurable by SFLC were excluded.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Part 2: Carfilzomib 20/27 mg/m²: Participants not previously treated with bortezomib received carfilzomib 20 mg/m² IV on Days 1, 2, 8, 9, 15, and 16 of Cycle 1. If all doses were well-tolerated the dose was escalated to 27 mg/m² IV on Days 1, 2, 8, 9, 15, and 16 for subsequent cycles, for up to 12 cycles.
Arm/Group | Part 1: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20/27 mg/m²
Number analyzed (Participants) | 31 | 53 | 66
percentage of participants | 16.1 [5.45 to 33.73] | 39.6 [26.5 to 54.0] | 53.0 [40.3 to 65.4]

2. Secondary Outcome: Best Overall Response Rate (ORR) in the Response Evaluable Population
Description: as for outcome 1
Time Frame: Disease response was assessed on Day 15 of Cycle 1, Day 1 of Cycles 2 through 12, End of Study, 30 days after last dose; median duration of treatment was 100 days for Part 1 and 170 days for Part 2 participants.
Population: The Response Evaluable population consists of all treated patients with measurable disease at Baseline as assessed by M-protein, SFLC or by quantitative serum Ig for certain patients with IgA myeloma, and with a baseline and at least 1 post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20/27 mg/m²
Number analyzed (Participants) | 35 | 59 | 67
percentage of participants | 17.1 [6.56 to 33.65] | 42.4 [29.6 to 55.9] | 52.2 [39.7 to 64.6]

3. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: Clinical Benefit Rate is defined as the percentage of participants with a best overall response of minimal response (MR) or better, i.e., a best overall response of sCR, CR, VGPR, PR, or MR. MR was defined as outlined by European Group for Blood and Marrow Transplantation (EBMT) criteria, defined as reduction of M-protein in serum of 25% to 49% and in urine of 50% to 89%, maintained for 6 weeks.
Time Frame: as for outcome 1
Population: Response Evaluable Population
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part 1: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20/27 mg/m²
Number analyzed (Participants) | 35 | 59 | 67
percentage of participants | 31.4 [16.85 to 49.29] | 59.3 [45.7 to 71.9] | 64.2 [51.5 to 75.5]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time from first evidence of PR or better to disease progression assessed by the IRC or death due to any cause. Patients lost to follow-up prior to disease progression or who were alive without disease progression before the analysis cutoff date were censored at the last disease assessment.
  Progressive disease was defined as any of the following:
  * An increase of M-protein in serum (absolute increase ≥ 0.5 g/dL) or urine (absolute increase ≥ 200 mg/24 hours) of > 25% from the nadir (if not zero).
  * Percentage of plasma cells in bone marrow ≥ 10%.
  * New or increased size of bone lesions or new plasmacytomas.
  * Patients without measurable serum and urine M-protein: 25% increase from nadir in the difference between involved and uninvolved FLC levels and absolute increase >10 mg/dL.
  * Development of hypercalcemia (corrected serum calcium > 11.5 mg/dL) attributed solely to the proliferative disorder.
  Median DOR was estimated using Kaplan-Meier methods.
Time Frame: Patients were followed for up to 2 years after study discontinuation. The data cutoff for the analysis is 30 November 2010 for Part 1 and 22 April 2011 for Part 2.
Population: Response Evaluable Population with a response of PR or better.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20/27 mg/m²
Number analyzed (Participants) | 6 | 25 | 35
months | NA [10.6 to NA] — Could not be estimated due to the low number of events | 13.1 [7.2 to NA] — Could not be estimated due to the low number of events | NA [NA to NA] — Could not be estimated due to the low number of events

5. Secondary Outcome: Time to Progression (TTP)
Description: Time to Progression is defined as the time from the start of treatment to IRC-determined disease progression. Patients who were lost to follow-up prior to documentation of disease progression, or who died before documentation of disease progression or who were alive and did not have documentation of disease progression before the data analysis cut-off date were censored at the last disease assessment.
  Median TTP was estimated using the Kaplan-Meier method.
Time Frame: Patients were followed for up to 2 years after study discontinuation. The data cutoff for the analysis is 30 November 2010 for Part 1 and 22 April 2011 for Part 2. Median follow-up time was 13.4 months for Part 1 and 11.5 months in Part 2.
Population: Response Evaluable Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20/27 mg/m²
Number analyzed (Participants) | 35 | 59 | 67
months | 4.6 [1.9 to 11.1] | 8.3 [6.0 to 12.3] | NA [11.3 to NA] — Could not be estimated due to the low number of events

6. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free Survival (PFS) is defined as the time from start of treatment to IRC determined disease progression or death due to any cause. Patients who were lost to follow-up prior to documentation of disease progression and patients who were alive without disease progression before a data analysis cut-off date were censored at the last disease assessment.
  Median PFS was estimated using the Kaplan-Meier method.
Time Frame: as for outcome 5
Population: Response Evaluable Population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20/27 mg/m²
Number analyzed (Participants) | 35 | 59 | 67
months | 4.6 [2.1 to 11.1] | 8.2 [6.0 to 12.3] | NA [11.3 to NA] — Could not be estimated due to the low number of events

7. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival is defined as the time from the start of study treatment to date of death due to any cause.
  Patients who were alive or lost to follow-up as of the data analysis cut-off date for the final OS analysis were censored at the date the patient was last known to be alive. Median OS was estimated using the Kaplan-Meier method.
Time Frame: Patients were followed for up to 2 years after study discontinuation. The data cutoff for the analysis is 19 November 2012 for Part 1 and 07 January 2013 for Part 2. Median follow-up time was 19.1 months for Part 1 and 35.9 months in Part 2.
Population: Safety Population includes all patients enrolled on study and who received at least 1 dose of carfilzomib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Part 1: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20/27 mg/m²
Number analyzed (Participants) | 35 | 59 | 70
months | 45.6 [28.4 to NA] — Could not be estimated due to the low number of events | NA [33.4 to NA] — Could not be estimated due to the low number of events | 37.3 [27.1 to NA] — Could not be estimated due to the low number of events

ADVERSE EVENTS:
Time Frame: From the first dose of study medication until 30 days after the last dose or initiation of new, non-protocol therapy for MM, whichever was first; median duration of treatment was 100 days for Part 1 and 170 days for Part 2 participants.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Part 1: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20 mg/m² | Part 2: Carfilzomib 20/27 mg/m²
Serious Adverse Events (participants affected / at risk) | 12/35 | 18/59 | 27/70
Other Adverse Events (participants affected / at risk) | 35/35 | 59/59 | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Carfilzomib 20 mg/m² (N=35) | Part 2: Carfilzomib 20 mg/m² (N=59) | Part 2: Carfilzomib 20/27 mg/m² (N=70)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1 | 0
Cardiac disorder (Cardiac disorders) | 0 | 0 | 1
Cardiac failure (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 2 | 2
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Disease progression (General disorders) | 1 | 1 | 1
Face oedema (General disorders) | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 1 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 2 | 1 | 3
Clostridium colitis (Infections and infestations) | 1 | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 1 | 0
Epiglottitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 3 | 6 | 6
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1
Pneumonia haemophilus (Infections and infestations) | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1 | 0
Sinusitis bacterial (Infections and infestations) | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Bone lesion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 2 | 3
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Haematoma (Vascular disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: Carfilzomib 20 mg/m² (N=35) | Part 2: Carfilzomib 20 mg/m² (N=59) | Part 2: Carfilzomib 20/27 mg/m² (N=70)
Anaemia (Blood and lymphatic system disorders) | 12 | 27 | 25
Leukopenia (Blood and lymphatic system disorders) | 6 | 12 | 4
Lymphopenia (Blood and lymphatic system disorders) | 6 | 20 | 13
Neutropenia (Blood and lymphatic system disorders) | 9 | 18 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 11 | 20 | 19
Bradycardia (Cardiac disorders) | 1 | 3 | 0
Tachycardia (Cardiac disorders) | 2 | 1 | 3
Tinnitus (Ear and labyrinth disorders) | 2 | 0 | 1
Diplopia (Eye disorders) | 2 | 1 | 1
Eye irritation (Eye disorders) | 3 | 1 | 3
Lacrimation increased (Eye disorders) | 1 | 4 | 1
Vision blurred (Eye disorders) | 3 | 6 | 4
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 5
Abdominal distension (Gastrointestinal disorders) | 3 | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 5 | 6 | 6
Bowel sounds abnormal (Gastrointestinal disorders) | 2 | 1 | 0
Constipation (Gastrointestinal disorders) | 8 | 15 | 10
Diarrhoea (Gastrointestinal disorders) | 13 | 21 | 18
Dyspepsia (Gastrointestinal disorders) | 3 | 4 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 3 | 1
Mouth ulceration (Gastrointestinal disorders) | 1 | 4 | 2
Nausea (Gastrointestinal disorders) | 21 | 32 | 31
Vomiting (Gastrointestinal disorders) | 15 | 14 | 14
Asthenia (General disorders) | 8 | 6 | 8
Chills (General disorders) | 6 | 15 | 14
Fatigue (General disorders) | 22 | 42 | 38
Gait disturbance (General disorders) | 4 | 2 | 1
Infusion site pain (General disorders) | 2 | 8 | 8
Injection site irritation (General disorders) | 2 | 4 | 3
Non-cardiac chest pain (General disorders) | 1 | 1 | 4
Oedema (General disorders) | 0 | 3 | 1
Oedema peripheral (General disorders) | 5 | 17 | 18
Pain (General disorders) | 7 | 11 | 9
Pitting oedema (General disorders) | 2 | 1 | 2
Pyrexia (General disorders) | 8 | 21 | 22
Bronchitis (Infections and infestations) | 2 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 2 | 1
Herpes zoster (Infections and infestations) | 3 | 1 | 2
Influenza (Infections and infestations) | 2 | 4 | 2
Nasopharyngitis (Infections and infestations) | 2 | 9 | 11
Oral candidiasis (Infections and infestations) | 2 | 1 | 2
Respiratory tract infection (Infections and infestations) | 2 | 0 | 2
Sinusitis (Infections and infestations) | 3 | 2 | 4
Upper respiratory tract infection (Infections and infestations) | 11 | 20 | 20
Urinary tract infection (Infections and infestations) | 3 | 9 | 3
Alanine aminotransferase increased (Investigations) | 10 | 7 | 2
Aspartate aminotransferase increased (Investigations) | 7 | 10 | 11
Blood albumin decreased (Investigations) | 3 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 2 | 3 | 1
Blood bicarbonate decreased (Investigations) | 3 | 1 | 3
Blood calcium decreased (Investigations) | 2 | 0 | 0
Blood calcium increased (Investigations) | 3 | 2 | 2
Blood creatinine increased (Investigations) | 12 | 14 | 10
Blood glucose increased (Investigations) | 4 | 1 | 1
Blood magnesium decreased (Investigations) | 3 | 2 | 1
Blood magnesium increased (Investigations) | 3 | 2 | 0
Blood phosphorus decreased (Investigations) | 6 | 7 | 5
Blood potassium decreased (Investigations) | 2 | 3 | 0
Blood potassium increased (Investigations) | 2 | 3 | 1
Blood sodium decreased (Investigations) | 3 | 5 | 0
Blood uric acid increased (Investigations) | 4 | 7 | 3
Breath sounds abnormal (Investigations) | 4 | 4 | 0
Carbon dioxide decreased (Investigations) | 0 | 3 | 0
Vibration test abnormal (Investigations) | 0 | 3 | 0
Weight decreased (Investigations) | 3 | 2 | 1
Weight increased (Investigations) | 2 | 1 | 4
Anorexia (Metabolism and nutrition disorders) | 3 | 8 | 5
Decreased appetite (Metabolism and nutrition disorders) | 3 | 3 | 5
Dehydration (Metabolism and nutrition disorders) | 1 | 4 | 3
Fluid overload (Metabolism and nutrition disorders) | 3 | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 2 | 1 | 2
Hypercalcaemia (Metabolism and nutrition disorders) | 3 | 6 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 7 | 7
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 5 | 8
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 3 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 4
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 6 | 8
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2 | 2 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 3 | 3 | 3
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 3 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 6 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 7 | 6
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 3 | 7
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 2 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 15 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 5
Chest wall pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 5
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 6 | 18
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 8 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 9 | 13
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 3 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Shoulder pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 1
Areflexia (Nervous system disorders) | 0 | 3 | 0
Dizziness (Nervous system disorders) | 7 | 12 | 10
Headache (Nervous system disorders) | 9 | 19 | 23
Hypoaesthesia (Nervous system disorders) | 9 | 10 | 8
Hyporeflexia (Nervous system disorders) | 2 | 4 | 1
Memory impairment (Nervous system disorders) | 2 | 3 | 3
Neuropathy (Nervous system disorders) | 2 | 3 | 2
Neuropathy peripheral (Nervous system disorders) | 2 | 4 | 5
Paraesthesia (Nervous system disorders) | 4 | 7 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 2 | 6
Sinus headache (Nervous system disorders) | 2 | 2 | 0
Anxiety (Psychiatric disorders) | 2 | 5 | 3
Confusional state (Psychiatric disorders) | 2 | 2 | 2
Depression (Psychiatric disorders) | 3 | 2 | 2
Insomnia (Psychiatric disorders) | 7 | 11 | 18
Mental status changes (Psychiatric disorders) | 2 | 2 | 0
Dysuria (Renal and urinary disorders) | 4 | 2 | 4
Pollakiuria (Renal and urinary disorders) | 0 | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 23 | 21
Crackles lung (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 | 29 | 19
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 7
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 7
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 3
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 6
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 5 | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Erythema (Skin and subcutaneous tissue disorders) | 4 | 5 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 6 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 3 | 1
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 3 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 7 | 5
Rash (Skin and subcutaneous tissue disorders) | 3 | 7 | 5
Nasal sinus drainage (Surgical and medical procedures) | 2 | 4 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 3 | 1
Flushing (Vascular disorders) | 3 | 1 | 4
Hot flush (Vascular disorders) | 1 | 4 | 1
Hypertension (Vascular disorders) | 6 | 8 | 13
Hypotension (Vascular disorders) | 2 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After the study is completed and all case report forms have been sent to Sponsor, Institution shall have the right to publish or otherwise make public any data resulting from the study under this agreement after publication of a multi-center publication coordinated by Sponsor with respect to the data resulting from the study, or 12 months after the Study is completed at all participating sites if a multi-center publication is not submitted by Sponsor for publication within such 12 month period.